CLINICAL TRIAL: NCT00006046
Title: Phase I Study of Humanized 3S193 (Anti-Lewis-Y) Antibody in Patients With Advanced Colorectal Carcinoma
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Advanced Colorectal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: poor recruitment
Sponsor: Ludwig Institute for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068062; MSKCC-00005 (Other: Memorial Sloan-Kettering Cancer Center); LUD1999-007 (Other: Ludwig Institute for Cancer Research)
Record Dates: First submitted 2000-07-05; First posted 2003-05-21 (Estimated); Results first posted 2021-08-09 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Hu3S193 monoclonal antibody

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Hu3S193 10 mg/m2 (Experimental): Hu3S193 was administered weekly for 8 consecutive weeks. The antibody was diluted in physiologic saline containing 5% human serum albumin and infused intravenously at a maximum rate of 100 mg/hour. If patients were stable or responding, they were eligible to receive 8-week maintenance cycles of hu3S193 at 10 mg/m2 starting in week 10 and continuing until progression.
  Interventions: Biological: monoclonal antibody hu3S193
- Hu3S193 25 mg/m2 (Experimental): Hu3S193 was administered weekly for 8 consecutive weeks. The antibody was diluted in physiologic saline containing 5% human serum albumin and infused intravenously at a maximum rate of 100 mg/hour. If patients were stable or responding, they were eligible to receive 8-week maintenance cycles of hu3S193 at 10 mg/m2 starting in week 10 and continuing until progression.
  Interventions: Biological: monoclonal antibody hu3S193
- Hu3S193 50 mg/m2 (Experimental): Hu3S193 was administered weekly for 8 consecutive weeks. The antibody was diluted in physiologic saline containing 5% human serum albumin and infused intravenously at a maximum rate of 100 mg/hour. If patients were stable or responding, they were eligible to receive 8-week maintenance cycles of hu3S193 at 10 mg/m2 starting in week 10 and continuing until progression.
  Interventions: Biological: monoclonal antibody hu3S193
- Hu3S193 100 mg/m2 (Experimental): Hu3S193 was administered weekly for 8 consecutive weeks. The antibody was diluted in physiologic saline containing 5% human serum albumin and infused intravenously at a maximum rate of 100 mg/hour. If patients were stable or responding, they were eligible to receive 8-week maintenance cycles of hu3S193 at 10 mg/m2 starting in week 10 and continuing until progression.
  Interventions: Biological: monoclonal antibody hu3S193
- Hu3S193 200 mg/m2 (Experimental): Hu3S193 was administered weekly for 8 consecutive weeks. The antibody was diluted in physiologic saline containing 5% human serum albumin and infused intravenously at a maximum rate of 100 mg/hour. If patients were stable or responding, they were eligible to receive 8-week maintenance cycles of hu3S193 at 10 mg/m2 starting in week 10 and continuing until progression.
  Interventions: Biological: monoclonal antibody hu3S193

INTERVENTIONS:
Biological: monoclonal antibody hu3S193

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase I trial to study the effectiveness of monoclonal antibody therapy in treating patients who have advanced colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity, maximum tolerated dose, and pharmacokinetics of monoclonal antibody hu3S193 in patients with advanced colorectal carcinoma.
* Determine the immune response in these patients treated with this regimen.

OUTLINE: This is a dose escalation study.

Patients receive monoclonal antibody hu3S193 (mAb hu3S193) IV over 30 minutes to 4 hours weekly for 8 weeks followed by 2 weeks of rest. Patients with stable or responding disease at week 10 receive maintenance mAb hu3S193 weekly. Courses repeat every 8 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of mAb hu3S193 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 3 of 6 patients experience dose limiting toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven stage IV colorectal carcinoma.
* Failed or refused conventional chemotherapy.
* Lewis Y antigen present on more than 50% of tumor cells.
* Measurable or evaluable disease.
* No central nervous system (CNS) tumor involvement.
* Karnofsky 80-100%.
* Life expectancy: At least 6 weeks.
* Granulocyte count greater than 1,500/mm^3.
* Platelet count greater than 100,000/mm^3.
* Bilirubin no greater than 1.0 mg/dL.
* Prothrombin time less than 3 times upper limit of normal.
* Creatinine no greater than 1.4 mg/dL.
* Female patients of childbearing age and male patients must be asked to use effective contraception during the study.
* At least 4 weeks since other prior immunotherapy. Exclusion Criteria
* New York Heart Association class III or IV heart disease.
* Serious infection requiring antibiotics or other serious illness.
* Pregnancy or nursing.
* History of bleeding gastric ulcers or pancreatitis.
* Diabetes mellitus requiring insulin.
* Human antimouse antibodies (HAMA).
* No prior mouse monoclonal antibody or antibody fragments.
* Illness requiring the use of steroids or other anti-inflammatory agents.
* Positive anti-hu3S193 antibody (HAHA) titer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2000-07-12 (Actual); Primary Completion 2001-10-05 (Actual); Study Completion 2002-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sydney Welt, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seven patients were entered into the 10mg/m2 dose cohort. No patients were entered into the other cohorts as the study was terminated due to poor recruitment.
Period: Overall Study
Arm/Group | Hu3S193 10 mg/m2 | Hu3S193 25 mg/m2 | Hu3S193 50 mg/m2 | Hu3S193 100 mg/m2 | Hu3S193 200 mg/m2
Started | 7 | 0 | 0 | 0 | 0
Completed | 2 | 0 | 0 | 0 | 0
Not Completed | 5 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0 | 0 | 0
Not completed — Disease Progression | 2 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients entered into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Hu3S193 10 mg/m2 | Hu3S193 25 mg/m2 | Hu3S193 50 mg/m2 | Hu3S193 100 mg/m2 | Hu3S193 200 mg/m2 | Total
Number analyzed (Participants) | 7 | 0 | 0 | 0 | 0 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  |  |  |  | 0
  Between 18 and 65 years | 6 |  |  |  |  | 6
  >=65 years | 1 |  |  |  |  | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 |  |  |  |  | 4
  Male | 3 |  |  |  |  | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 |  |  |  |  | 2
  Not Hispanic or Latino | 5 |  |  |  |  | 5
  Unknown or Not Reported | 0 |  |  |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  |  |  | 0
  Asian | 0 |  |  |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  |  |  | 0
  Black or African American | 0 |  |  |  |  | 0
  White | 7 |  |  |  |  | 7
  More than one race | 0 |  |  |  |  | 0
  Unknown or Not Reported | 0 |  |  |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 |  |  |  |  | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose-limiting Toxicities (DLTs)
Description: Toxicity was graded in accordance with the Common Toxicity Scale developed by NCI (1998) where Grade 1 represents the lowest toxicity grade and Grade 5 death. Dose-limiting toxicity (DLT) was defined as Grade 3 and Grade 4 adverse events which were at least possibly related to study treatment.
Time Frame: up to 10 weeks.
Population: All patients who entered the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Hu3S193 10 mg/m2 | Hu3S193 25 mg/m2 | Hu3S193 50 mg/m2 | Hu3S193 100 mg/m2 | Hu3S193 200 mg/m2
Number analyzed (Participants) | 7 | 0 | 0 | 0 | 0
Participants | 1 | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Patients With Tumor Responses
Description: Complete response (CR); disappearance of all measurable disease lasting a minimum of 4 weeks. Partial Response (PR); 50% or greater decrease in the sum of the products of the perpendicular diameters or all measurable lesions, without development of new lesions or increase in size of any lesion, lasting a minimum of 4 weeks. Progressive disease (PD); Appearance of new lesions or increase by 25% or more in size of any measurable lesion. Stable disease (SD); Not meeting criteria for response or progression.
Time Frame: 8 weeks
Population: All patients who entered the study and had tumor assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Hu3S193 10 mg/m2 | Hu3S193 25 mg/m2 | Hu3S193 50 mg/m2 | Hu3S193 100 mg/m2 | Hu3S193 200 mg/m2
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Participants
  CR | 0 | 0 | 0 | 0 | 0
  PR | 0 | 0 | 0 | 0 | 0
  SD | 0 | 0 | 0 | 0 | 0
  PD | 4 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 10 weeks
Description: Adverse Events (AEs) were collected on the adverse event page of the Case Report Form (CRF). AEs were graded in accordance with the Common Toxicity Scale developed by NCI (1998).
  Seven patients were entered into the 10 mg/m2 dose cohort. No patients were entered into the other cohorts as the study was terminated due to poor recruitment.
Arm/Group | Hu3S193 10 mg/m2 | Hu3S193 25 mg/m2 | Hu3S193 50 mg/m2 | Hu3S193 100 mg/m2 | Hu3S193 200 mg/m2
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 5/7 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 3/7 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hu3S193 10 mg/m2 (N=7) | Hu3S193 25 mg/m2 (N=0) | Hu3S193 50 mg/m2 (N=0) | Hu3S193 100 mg/m2 (N=0) | Hu3S193 200 mg/m2 (N=0)
Actinomycosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hu3S193 10 mg/m2 (N=7) | Hu3S193 25 mg/m2 (N=0) | Hu3S193 50 mg/m2 (N=0) | Hu3S193 100 mg/m2 (N=0) | Hu3S193 200 mg/m2 (N=0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Chills (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No